CLINICAL TRIAL: NCT00996593
Title: Phase II Study of Iodine-131 Anti-B1 Antibody for Non Hodgkin's Lymphoma Patients Who Have Previously Received Rituximab
Brief Title: Study of Iodine-131 Anti-B1 Antibody for Patients With Non Hodgkin's Lymphoma Who Have Previously Received Rituximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104507
Record Dates: First submitted 2009-10-08; First posted 2009-10-16 (Estimated); Results first posted 2012-01-26 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-10

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Tositumomab; radioimmunotherapy; rituximab; anti-B1; I 131; Bexxar; iodine; non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

ARMS (1):
- open-label, single arm (Experimental)
  Interventions: Biological: Anti-B1 Antibody and Iodine-131 Anti-B1 Antibody (Tositumomab and Iodine I 131 Tositumomab)

INTERVENTIONS:
Biological: Anti-B1 Antibody and Iodine-131 Anti-B1 Antibody (Tositumomab and Iodine I 131 Tositumomab) — Patients will receive an infusion of unlabeled Anti-B1 Antibody (450 mg) followed by an infusion of Anti-B1 Antibody (35 mg) containing 5 mCi of Iodine-131 (dosimetric dose). Whole body gamma camera scans will be obtained on Day 0; Day 2, 3, or 4; and Day 6 or 7 following the dosimetric dose. Patients will then receive an infusion of unlabeled Anti-B1 Antibody (450 mg) followed by an infusion of 35 mg Anti-B1 Antibody containing a patient-specific dose of Iodine-131 calculated to deliver a 75 cGy total body radiation dose (therapeutic dose). Patients who have platelet counts of 100,001-149,999 cells/mm3 will receive 65 cGy; obese patients will be dosed based upon 137% of their lean body mass. Patients will be treated with a thyroid blocking agent 24 hours prior to the dosimetric dose and continuing for 14 days following the therapeutic dose.

SUMMARY:
This is a single-arm, open-label, multicenter study of Iodine I-131 Anti B1 Antibody (Tositumomab and Iodine I 131 Tositumomab) for treatment of non-Hodgkin's lymphoma (NHL) who were previously treated with rituximab antibody. Patients must have been treated with at least 4 doses of rituximab and have progressed during or following rituximab therapy.

Patients will undergo two dosing phases of study. In the first phase, termed the "dosimetric dose", patients will receive an infusion of unlabeled Anti-B1 Antibody (450 mg) over 70 minutes immediately followed by a 30-minute infusion of Anti-B1 Antibody (35 mg) which has been radiolabeled with 5 mCi of Iodine-131. Whole body gamma camera scans will be obtained on Day 0; Day 2, 3, or 4; and Day 6 or 7 following the dosimetric dose. Using the dosimetric data from three imaging timepoints, a patient-specific dose of Iodine-131 will be calculated to deliver the desired total body dose of radiotherapy. In the second phase, termed the "therapeutic dose", patients will receive a 70-minute infusion of unlabeled Anti-B1 Antibody (450 mg) immediately followed by a 30-minute infusion of 35 mg Anti-B1 Antibody labeled with a patient-specific dose of Iodine-131 to deliver a whole body dose of 75 cGy to patients with no hematologic risk factors. Patients who have platelet counts of 100,001-149,999 cells/mm3 will receive 65 cGy and patients who are obese will be dosed based upon 137% of their lean body mass. Patients will be treated with either saturated solution potassium iodide (SSKI), Lugol's solution, or potassium iodide tablets starting at least 24 hours prior to the first infusion of the Iodine-131 Anti-B1 Antibody (i.e., dosimetric dose) and continuing for 14 days following the last infusion of Iodine-131 Anti-B1 Antibody (i.e., therapeutic dose).

The endpoints of the study are to determine the response rate, complete response rate, duration of response, and time to progression or death, based on both a Masked Independent Randomized Radiographic and Oncologic Review (MIRROR) panel and the Investigators, and the Investigators' assessment of safety and survival of survival of Iodine-131 Anti-B1 Antibody therapy in NHL patients who have previously been treated with rituximab.

ELIGIBILITY:
Inclusion Criteria

* Patients must have a histologically confirmed diagnosis of low-grade non-Hodgkin's B-cell lymphoma according to International Working Formulation.
* Patients must have evidence that their tumor tissue expresses the CD20 antigen. Immunoperoxidase stains of paraffin-embedded tissue showing positive reactivity with L26 antibody or immunoperoxidase stains of frozen tissue showing positive reactivity with Anti-B1 Antibody or evidence of CD20 positivity by flow cytometry are acceptable evidence of CD20 positivity.
* Patients must have been treated with at least 4 doses of rituximab at any time and failed to achieve an objective response (CR, CCR, PR) or relapse/progressed during treatment or following the completion of rituximab therapy.
* Patients must have a performance status of at least 60% on the Karnofsky Scale and an anticipated survival of at least 3 months.
* Patients must have an absolute granulocyte count >1500 cells/mm3 (US) and a platelet count >100,000 cells/mm3 (US) within 14 days of study entry. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
* Patients must have adequate renal function (defined as serum creatinine <1.5 x upper limit of normal [ULN]) and hepatic function (defined as total bilirubin <1.5 x ULN and aspartate transaminase [AST] <5 x ULN) within 14 days of study entry.
* Patients must have bi-dimensionally measurable disease. At least one lesion must be greater than or equal to 2 x 2 cm (by computed tomography [CT] scan).
* Patients must be at least 18 years of age.
* Patients must give written informed consent and sign an IRB/EC- approved informed consent form prior to study entry.

Exclusion Criteria

* Patients with more than an average of 25% of the intratrabecular marrow space involved by lymphoma in bone marrow biopsy specimens as assessed microscopically within 42 days of study entry. Bilateral posterior iliac crest core biopsies are required if the percentage of intratrabecular space involved exceeds 10% on a unilateral biopsy. The mean of bilateral biopsies must be no more than 25%.
* Patients who received cytotoxic chemotherapy, radiation therapy, immunosuppressants, or cytokine treatment within 4 weeks prior to study entry (6 weeks of nitrosourea compounds) or who exhibit persistent clinical evidence of toxicity. The use of systemic steroids must be discontinued at least 1 week prior to study entry.
* Patients with prior hematopoietic stem cell transplant following high-dose chemotherapy or chemo/radiotherapy.
* Patients with active obstructive hydronephrosis.
* Patients with evidence of active infection requiring intravenous (IV) antibiotics at the time of study entry.
* Patients with New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation.
* Patients with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years.
* Patients with known HIV infection.
* Patients with known brain or leptomeningeal metastases.
* Patients who are pregnant or nursing. Patients of childbearing potential must undergo a pregnancy test within 7 days of study entry and radiolabeled antibody is not to be administered until a negative result is obtained. Males and females must agree to use effective contraception for 6 months following the radioimmunotherapy.
* Patients with previous allergic reactions to iodine. This does not include reacting to IV iodine-containing contrast materials.
* Patients who previously received radioimmunotherapy.
* Patients with progressive disease within 1 year of irradiation arising in a field that has been previously irradiated with > 3500 cGy.
* Patients who are HAMA positive.
* Patients who are concurrently receiving either approved or non-approved (through another protocol) anti-cancer drugs or biologics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 1998-07; Primary Completion 2001-04 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: GSK Clinical Study Register — http://www.gsk-clinicalstudyregister.com/result_detail.jsp?protocolId=CP-97-012&studyId=2951&compound=Tositumomab
- Available data/document: Individual Participant Data Set: 104507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104507 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received radioimmunotherapy of tositumomab (TST) and Iodine I 131 TST in 2 phases: Phase 1, dosimetric dose; Phase 2, therapeutic dose. After radioimmunotherapy, participants could have entered a 10-year Long-Term Follow-Up study (Study BEX104526; NCT00240591) for continued evaluation.
Groups:
- TST and Iodine I 131 TST: Participants received a dosimetric dose (DD) consisting of 450 milligrams (mg) of tositumomab (TST) intravenously (IV) followed by 5.0 millicurie (mCi) of Iodine I 131 and 35 mg of TST IV. The therapeutic dose (TD) consisting of 450 mg of TST IV, followed by a participant-specific dose of I 131 (75 centigray [cGy] or 65 cGy) and 35 mg of TST IV, was administered 7-14 days after the DD. Participants who had completed at least 2 years of follow-up after administration of TST/I 131 TST during the TD phase and had signed the informed consent to participate in the Long-Term Follow-Up (LTFU) study (BEX104526) were followed for up to 10 years. Participants did not receive any study medication during the LTFU study.
Period: Dosimetric and Therapeutic Treatment
Arm/Group | TST and Iodine I 131 TST
Started | 43
Completed | 0
Not Completed | 43
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 3
Not completed — Progressive Disease | 22
Not completed — Death | 1
Not completed — Enrolled in BEX104526 | 6
Not completed — Did Not Receive Any Study Drug | 3
Not completed — Non-compliance | 1
Period: Long-Term Follow-Up
Arm/Group | TST and Iodine I 131 TST
Started | 9 (9 of the 40 participants withdrawing from Study BEX104507 enrolled in long-term follow-up study.)
Completed | 6
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Site Closed | 1

BASELINE CHARACTERISTICS:
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics are summarized for the Intent-to-Treat (ITT) Population, comprised of all participants who were enrolled into the study and received at least one dose of study drug.
  Years | 57.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics are summarized for the Intent-to-Treat (ITT) Population, comprised of all participants who were enrolled into the study and received at least one dose of study drug.
  Participants
    Female | 13
    Male | 27
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics are summarized for the Intent-to-Treat (ITT) Population, comprised of all participants who were enrolled into the study and received at least one dose of study drug.
  participants
    White | 33
    Hispanic | 3
    Asian | 1
    Black | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) With Confirmed Response as Assessed by the Investigator
Description: Responses had to be confirmed by 2 separate evaluations occurring >=4 weeks apart. Par. with confirmed response include those with Complete Response (CR: complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease), Clinical Complete Response (CCR: complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present), or Partial Response (PR: >=50% reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions; no new lesions).
Time Frame: Participants were evaluated until death (up to 80.2 months in Study BEX104507) or were followed in the long-term follow-up study for up to 10.5 years
Population: Intent-to-Treat (ITT) Exposed Population: all participants who were enrolled into the study and received at least one dose of study drug. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 34
participants | 26
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; Percentage of participants = 65, 95% CI 2-sided [50 to 80] — The estimated value represents the percentage of participants with complete response

2. Primary Outcome: Number of Participants With Confirmed Complete Response (CR) as Assessed by the Investigator
Description: CR is defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for confirmed response were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 34
participants | 9
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; Percentage of participants = 23, 95% CI 2-sided [10 to 35] — The estimated value represents the percentage of participants with complete response

3. Primary Outcome: Number of Participants With Confirmed Complete Response Plus Clinical Complete Response (CR + CCR) as Assessed by the Investigator
Description: CCR is defined as the complete resolution of all disease-related symptoms; residual foci, thought to be residual scar tissue, are present. Generally, an unchanging lesion =<2 centimeters (cm) in diameter by radiographic evaluation or =<1 cm in diameter by physical examination can be considered scar tissue. The extent of disease must be unchanged or decreased upon follow-up evaluations. If the extent of disease was unchanged or if further decreases occurred for 6 months or longer, the participant was reclassified as having a CR.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for CR + CCR were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 34
participants | 15
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; Percentage of participants = 38, 95% CI 2-sided [22 to 53] — The estimated value represents the percentage of participants with complete response

4. Primary Outcome: Number of Participants With Confirmed Partial Response (PR) as Assessed by the Investigator
Description: Confirmed PR is defined as a >=50 percent reduction in the sum of the products of the longest perpendicular diameters of all measurable lesions, with no new lesions.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants evaluable for confirmed PR were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 34
participants | 11
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; Percentage of participants = 28, 95% CI 2-sided [14 to 41] — The estimated value represents the percentage of participants with complete response

5. Primary Outcome: Duration of Response for All Confirmed Responders (CR, CCR, or PR) as Assessed by the Investigator
Description: Response duration is defined as the time from the first documented response until disease progression.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants with confirmed response and those who experienced progressive disease were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 16
months | 22.2 [14.9 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval.

6. Primary Outcome: Duration of Response for Confirmed CR as Assessed by the Investigator
Description: Response duration is defined as the time from the first documented response until disease progression. Disease progression is defined as a >=25% increase from the nadir value of the sum of the products of the longest perpendicular diameters of all measureable lesions or the appearance of any new lesion. Individual lesions must be >2 centimeters (cm) in diameter by radiographic evaluation or >1 cm in diameter by physical examination.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants with confirmed CR and those who experienced progressive disease were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 4
months | NA [NA to NA] — The median (50% quartile) was not reached/calculated/available because there were not enough events to reach a median on the Kaplan Meier curve.

7. Primary Outcome: Duration of Response for CR and CCR as Assessed by the Investigator
Description: Response duration is defined as the time from the first documented response until disease progression.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants with confirmed CR + CCR response and those who experienced progressive disease were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 6
months | NA [NA to NA] — The median (50% quartile) was not reached/calculated/available because there were not enough events to reach a median on the Kaplan Meier curve.

8. Primary Outcome: Duration of Response for All Confirmed Partial Responders as Assessed by the Investigator
Description: Response duration is defined as the time from the first documented response until progressive disease.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants with confirmed PR and those who experienced progressive disease were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 10
months | 8.8 [4.4 to 15.9]

9. Primary Outcome: Number of Participants With or Without (w/o) a Prior Response to Rituximab (Before Entry Into This Study) Who Were Classified as Responders in This Study
Description: Response corresponds to the best response evaluation (ordered by CR, CCR, and PR) and does not require subsequent confirmation. Participants with CR, CCR, or PR are considered to be responders. A prior response to rituximab refers to a CR, CCR, or PR after rituximab treatment before enrollment into Study BEX104507.
Time Frame: as for outcome 1
Population: Subset of ITT Exposed Population. Only those participants who had received rituximab prior to entry into this study were evaluated.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
participants
  Responders with prior response to Rituximab; n=16 | 12
  Responders w/o prior response to Rituximab; n=24 | 16
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; p = 1.0, Fisher Exact — With prior response; Percentage of responders = 75, 95% CI 2-sided [54 to 96] — The estimated value represents the percentage of participants with response
Statistical Analysis 2: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; p = 1.0, Fisher Exact — Without prior response; Percentage of responders = 70, 95% CI 2-sided [51 to 88] — The estimated value represents the percentage of participants with response

10. Primary Outcome: Duration of Response for All Participants Classified as Responders With or Without a Prior Response to Rituximab
Description: Duration of response is defined as the time from the first documented response to disease progression.
Time Frame: as for outcome 1
Population: Subset of ITT Exposed Population. Only those participants who had received rituximab prior to entry into this study were evaluated. Only those participants with a response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 28
months
  Responders with prior response to Rituximab; n=12 | 18.6 [7.2 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval.
  Responders w/o prior response to Rituximab; n=16 | 19.2 [8.8 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval.
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; p = 0.8, Fisher Exact

11. Primary Outcome: Number of Participants With or Without (w/o) a Prior Response to Rituximab (Before Entry Into This Study) Who Were Classified as Having a Complete Response (CR) in This Study
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
participants
  Responders with prior response to Rituximab; n=16 | 5
  Responders w/o prior response to Rituximab; n=24 | 4
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; p = 1.0, Fisher Exact — With prior response; Percentage of responders = 31, 95% CI 2-sided [9 to 54] — The estimated value represents the percentage of participants with response
Statistical Analysis 2: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; p = 1.0, Fisher Exact — Without prior response; Percentage of responders = 17, 95% CI 2-sided [2 to 33] — The estimated value represents the percentage of participants with response

12. Primary Outcome: Duration of Response for All Participants With CR With or Without a Prior Response to Rituximab
Description: Duration of response is defined as the time from the first documented response to disease progression.
Time Frame: as for outcome 1
Population: Subset of ITT Exposed Population. Only those participants who had received rituximab prior to entry into this study were evaluated. Only those participants with confirmed response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 9
months
  Responders with prior response to Rituximab; n=5 | 47.3 [4.2 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval.
  Responders w/o prior response to Rituximab; n=4 | NA [NA to NA] — The median (50% quartile) was not reached/calculated/available because there were not enough events to reach a median on the Kaplan Meier curve.
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; p = 0.2, Fisher Exact

13. Primary Outcome: Progression-free Survival for Participants With or Without a Prior Response to Rituximab
Description: Progression-free survival is defined as the time from treatment start to the first documented occurrence of disease progression or death.
Time Frame: as for outcome 1
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 9
months
  Responders with prior response to Rituximab; n=5 | 13.0 [3.3 to 49.1]
  Responders w/o prior response to Rituximab; n=4 | 8.9 [5.1 to 25.6]
Statistical Analysis 1: Comparison: TST and Iodine I 131 TST; Test type: Superiority or Other; p = 0.9, Log Rank

14. Primary Outcome: Time to Progression of Disease or Death in All Responders, Participants With CR + CCR, and Participants With PR as Assessed by the Investigator
Description: Progression-free survival or time to progression is defined as the time from the dosimetric dose to the first documented occurrence of disease progression or death.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who experienced progression were evaluated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 30
months
  All responders, n=30 | 10.4 [5.7 to 18.6]
  CR + CCR, n=15 | NA [NA to NA] — The median (50% quartile) was not reached/calculated/available because there were not enough events to reach a median on the Kaplan Meier curve.
  PR, n=11 | 9.2 [5.7 to 17.7]

15. Secondary Outcome: Number of Participants With the Indicated Adverse Events (AE) Possibly or Probably Related to Study Drug and Experienced by at Least 5% of Participants
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The Investigator assessed whether the adverse event was possibly or probably related to study drug. In addition, all laboratory-derived hematologic toxicities were assumed to be possibly or probably related to study drug.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
participants
  Absolute Neutrophil Count (ANC) <1000 cells/cm^3 | 16
  White Blood Cells (WBC) <2000 cells/cm^3 | 15
  Platelets <50000 cells/cm^3 | 10
  Hemoglobin <8.0 grams/deciliter (g/dL) | 5
  Pyrexia | 9
  Fatigue | 7
  Chills | 4
  Edema Peripheral | 3
  Asthenia | 2
  Malaise | 2
  Arthralgia | 5
  Myalgia | 3
  Nausea | 7
  Vomiting | 5
  Anaemia | 4
  Thrombocytopenia | 3
  Neutropenia | 2
  Pruritus | 3
  Rash | 3
  Epistaxis | 3
  Productive Cough | 2
  Decreased Appetite | 2
  Upper Respiratory Tract Infection | 3
  Myelodysplastic Syndrome/ Acute Myeloid Leukemia | 2
  Headache | 3

16. Secondary Outcome: Number of Participants With the Indicated Type of Infection
Description: An infection is the colonization of a host organism by a parasite species. Infecting parasites seek to use the host's resources to reproduce, often resulting in disease. Specimen samples of the body fluid are cultured for testing whether the infectious organism is present and grown in the culture media to assess the growth pattern of the organisms present in the specimen. The culture results could be positive or negative. The positive culture results indicate that the tested participant has the infection under investigation, in which case therapeutic treatment with anti-infective is required.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
participants
  Any Infection; n=40 | 22
  No Infection; n=40 | 18
  Meningitis; n=22 | 0
  Pyelonephritis; n=22 | 0
  Sepsis; n=22 | 1
  Pneumonia; n=22 | 5
  Endocarditis/ Pericarditis; n=22 | 0
  Peritonitis; n=22 | 0
  Other Infections; n=22 | 17

17. Secondary Outcome: Number of Participants With an Infection for Which Anti-infectives Were Administered
Description: Anti-infectives are capable of acting against infection, by inhibiting the spread of an infectious agent or by killing the infectious agent outright. Anti-infective is a general term that encompasses antibacterials, antibiotics, antifungals, antiprotozoans, and antivirals.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who had infection during the study and during the follow-up period were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 22
participants
  Anti-infective Administered | 19
  Anti-infective Not Administered | 3

18. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE) Related to Study Drug
Description: An SAE is any event occurring at any dose that results in any of the following: death, a life-threatening adverse drug experience (ADE; at immediate risk of death from the experience as it occurred), inpatient hospitalization/prolongation of existing hospitalization, a persistent/significant disability/incapacity, or a congenital anomaly/birth defect. Medical events that may not result in death, be life-threatening, or require hospitalization may be considered to be a serious ADEs when based upon appropriate medical judgment. Relatedness was based on the investigator's medical judgement.
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants who experienced any SAE were analyzed.
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 13
participants
  Myelodysplastic syndrome/Acute myeloid leukemia | 2
  Malignant hepatobiliary neoplasm | 1
  Squamous cell carcinoma | 1
  Tumor lysis syndrome | 1
  Pyrexia | 1
  Anemia | 1

19. Secondary Outcome: Time to Nadir and Time to Recovery to Baseline in Hematologic Laboratory Evaluations
Description: Nadir is defined as the lowest laboratory value recorded following the administration of the study medication. Time to recovery to baseline in hematologic laboratory evaluations is the time required for recovery from nadir values to baseline values.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Median (Full Range); unit: days
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
days
  Time to nadir ANC, n=40 | 43.5 [3 to 90]
  Time to nadir hemoglobin, n=40 | 43 [3 to 88]
  Time to nadir platelets, n=40 | 34.5 [3 to 58]
  Time to nadir WBC count, n=40 | 43 [3 to 90]
  Time to recovery to baseline ANC, n=32 | 71 [58 to 76]
  Time to recovery to baseline hemoglobin, n=29 | 74 [43 to 83]
  Time to recovery to baseline platelets, n=29 | 55 [50 to 71]
  Time to recovery to baseline WBC count, n=28 | 78 [71 to 85]

20. Secondary Outcome: Nadir Values for ANC, a Hematologic Parameter
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. ANC is a measure of the number of neutrophil granulocytes present in the blood. Neutrophils are a type of white blood cell that fights against infection.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Median (Full Range); unit: cells/millimeters cubed (mm^3)
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
cells/millimeters cubed (mm^3) | 1.2 [0 to 6]

21. Secondary Outcome: Nadir Values for Hemoglobin, a Hematologic Parameter
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. Hemoglobin is the iron-containing oxygen-transport metalloprotein in the red blood cells.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Median (Full Range); unit: G/dL
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
G/dL | 11 [7 to 14]

22. Secondary Outcome: Nadir Values for Hematologic Parameters Platelets and WBC Count
Description: Nadir is defined as the lowest laboratory value recorded following the administration of study medication. Platelets and WBCs are types of blood cells.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Median (Full Range); unit: cells/microliter
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
cells/microliter
  Platelets (10000 cells/microliter) | 84.5 [9 to 168]
  WBC count (1000 cells/microliter) | 2.3 [1 to 7]

23. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 Hematologic Toxicities
Description: Adverse events were graded using the Common Toxicity Criteria from the Cancer Therapy Evaluation Program, Division of Cancer Therapy, National Cancer Institute. Grades: 0 = No adverse event or within normal limits; 1 = Mild adverse event; 2 = Moderate adverse event; 3 = Severe and undesirable adverse event; 4 = Life-threatening or disabling adverse event; 5 = Death related to adverse event.
Time Frame: as for outcome 1
Population: ITT Exposed Population
Measure: Number; unit: participants
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
participants
  ANC | 16
  Hemoglobin | 5
  Platelets | 10
  WBC count | 15

24. Secondary Outcome: Duration of the Indicated Grade 3 or Grade 4 Hematologic Toxicities
Description: as for outcome 23
Time Frame: as for outcome 1
Population: ITT Exposed Population. All participants with Grade 3 or Grade 4 hematologic toxicities were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 40
days
  ANC, n=16 | 14 [7 to 327]
  Hemoglobin, n=5 | 28 [11 to 71]
  Platelets, n=10 | 25 [8 to 48]
  WBC count, n=15 | 11 [7 to 235]

25. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from the treatment start date to the date of death from any cause.
Time Frame: as for outcome 1
Population: ITT Exposed Population. Only those participants who died during the study and during the follow-up period were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TST and Iodine I 131 TST
Number analyzed (Participants) | 20
months | 80 [24.8 to NA] — The SAS procedure was not able to calculate the upper limit of the confidence interval.

ADVERSE EVENTS:
Time Frame: Participants were evaluated until death or were followed in the long-term follow-up study for up to 10.5 years.
Arm/Group | TST and Iodine I 131 TST
Serious Adverse Events (participants affected / at risk) | 13/40
Other Adverse Events (participants affected / at risk) | 37/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and Iodine I 131 TST (N=40)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Human anti-mouse antibody positive (Investigations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TST and Iodine I 131 TST (N=40)
Fatigue (General disorders) | 12
Pyrexia (General disorders) | 11
Chills (General disorders) | 4
Asthenia (General disorders) | 3
Oedema peripheral (General disorders) | 3
Malaise (General disorders) | 2
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Face oedema (General disorders) | 1
Ill-defined disorder (General disorders) | 1
Infusion site erythema (General disorders) | 1
Oedema (General disorders) | 1
Pain (General disorders) | 1
ANC <1000 cells/mm^3 (Blood and lymphatic system disorders) | 16
WBC < 2000 cells/mm^3 (Investigations) | 15
Platelets <50000 cells/mm^3 (Investigations) | 10
Hemoglobin <8.0 g/dL (Investigations) | 5
Upper respiratory tract infection (Infections and infestations) | 8
Pneumonia (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal mass (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hypovolaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Cardiac murmur (Investigations) | 2
Body temperature increased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Human anti-mouse antibody positive (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tachycardia (Cardiac disorders) | 3
Arrhythmia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Dissociation (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Hypotension (Vascular disorders) | 3
Deep vein thrombosis (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Conjunctivitis (Eye disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.